CLINICAL TRIAL: NCT06147037
Title: A Phase 1, First-in-human, Multicentre, Open-label, Dose Escalation Study of [225Ac]-FPI-2068 in Adult Patients With Advanced Solid Tumours
Brief Title: A Phase 1, Dose-escalation Study of [225Ac]-FPI-2068 in Adult Patients With Advanced Solid Tumours
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FPI-2068-101
Record Dates: First submitted 2023-11-20; First posted 2023-11-27 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumor; Metastatic Colorectal Carcinoma; Head and Neck Squamous Cell Carcinoma; Non-small Cell Lung Cancer; Pancreatic Ductal Adenocarcinoma; Gastric Cancer; Renal Cell Carcinoma
Keywords: FPI-2068; FPI-2107; FPI-2053; Actinium-225; 225Ac; Indium-111; 111In; Solid tumors; Targeted alpha therapy; TAT; Epidermal growth factor receptor; EGFR; Mesenchymal-epithelial transition factor; cMET; Bispecific antibody; Radioimmuno-SPECT agent; Radioimmuno-therapeutic agent; Monoclonal antibody; Bifunctional chelating agent; Radiopharmaceutical therapy; Alpha particle emitter; Directed bispecific monovalent antibody; bsAb; Bifunctional chelate; mCRC; HNSCC; NSCLC; PDAC; GC; RCC; RLT; Radioligand Therapy; EGFRm; EGFRwt
MeSH Terms: conditions — Colorectal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Exploration and Dose Escalation (Experimental): The study conducted in two parts: Part A Dose Exploration and Part B Dose Escalation
  FPI-2053 dose exploration to determine the optimal pre-dose administration of FPI-2053 with a fixed dose of [225Ac]-FPI-2068.
  [225Ac]-FPI-2068 dose escalation with the optimal dose of FPI-2053 as determined in Part A.
  Interventions: Drug: FPI-2053; Drug: [111In]-FPI-2107; Drug: [225Ac]-FPI-2068

INTERVENTIONS:
Drug: FPI-2053 — FPI-2053 is a bispecific antibody that targets EGFR and cMET
Drug: [111In]-FPI-2107 — [111In]-FPI-2107 is an imaging agent in which indium-111 is conjugated to FPI-2053.
  Participants will have a fixed dose of [111In]-FPI-2107 followed by imaging scans (with or without pre-administration of FPI-2053).
Drug: [225Ac]-FPI-2068 — [225Ac]-FPI-2068 is a radiopharmaceutical therapy in which an alpha emitter, actinium-225, is conjugated to FPI-2053.
  Participants will be dosed through IV administration every 56 days for up to 3 cycles of the Treatment Period.

SUMMARY:
This is a first-in-human, Phase 1, non-randomized, multicenter, open-label clinical study designed to investigate the safety, tolerability, dosimetry, biodistribution, and pharmacokinetics (PK) of [225Ac]-FPI-2068, [111In]-FPI-2107, and FPI-2053 in metastatic and/or recurrent solid tumors (HNSCC, NSCLC, mCRC, PDAC, GC, RCC).

DETAILED DESCRIPTION:
The study will be conducted in 2 parts:

Part A: optimization of the FPI-2053 dose (treatment with dose level 1 of [225Ac]-FPI-2068 - fixed dose).

Part B: dose escalation of [225Ac]-FPI-2068 with optimal FPI-2053. Part B will commence once the optimal dose of FPI-2053 is determined in Part A. The RP2D will be determined from Part B based on all available safety, efficacy, PK, and dosimetry information.

ELIGIBILITY:
Key Inclusion Criteria:

Histologically and/or cytologically confirmed solid tumor that is metastatic, locally advanced, recurrent or inoperable.

Disease that has progressed despite prior treatment, and for which additional effective standard therapy is not available or is contraindicated, not tolerable, or the participant refuses standard therapy.

Measurable disease as defined by RECIST Version 1.1

ECOG Performance status of 0 or 1

Adequate organ function

Key Exclusion Criteria:

Previous treatment with any systemic radiopharmaceutical

Prior anti-cancer therapy unless adequate washout and recovery from toxicities

Contraindications to or inability to perform the imaging procedures required in this study

Radiation therapy (RT) within 28 days prior to the first dose of [111In]-FPI-2107

Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (≥ once per month)

Patients with known CNS metastatic disease unless treated and stable

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2028-05-12 (Estimated); Study Completion 2028-05-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate safety and tolerability of [111In]-FPI-2107, FPI-2053, and [225Ac]-FPI-2068 | From informed consent up to approximately 5 years post last administration
  Frequency, duration, and severity of AEs, DLTs, and changes in clinical, laboratory, and ECG parameters compared to baseline
Determine radiation dose of [111In]-FPI-2107 and [225Ac]-FPI-2068 to whole body, organs, and selected regions of interest. | Within 56 days of administration
  Changes in uptake of [111In]-FPI-2107 and projected RAD of [225Ac]-FPI-2068 by imaging following the administration of varying doses of FPI-2053
Determine the RP2D of [225Ac]-FPI-2068, given with or without FPI-2053 | 56 days post administration
  Estimates of residence time and absorbed radiation doses to the whole body, organs, and selected regions of interest for [111In]-FPI-2107 and [225Ac]-FPI-2068.
Determine the effect of predose administration of varying doses of FPI-2053 on the radiation dosimetry of [111In]-FPI-2107 and [225Ac]-FPI-2068 to whole body, organs, and selected regions of interest. | 56 days post-administration
  Changes in uptake of [111In]-FPI- 2107 and projected RAD of [225Ac]-FPI-2068 by imaging following the administration of varying doses of FPI-2053

SECONDARY OUTCOMES:
Assess preliminary anti-tumor activity of [225Ac]-FPI-2068 | Approximately 5 years post final administration
  * Tumor assessments will be based on RECIST v1.1 (Eisenhauer et al, 2009) and will be performed every 8 weeks (± 1 weeks) after first [225Ac]-FPI-2068 dose. During Long term follow up will be every 3 months (± 2 weeks) for 2 years and then every 6 months for 3 years, or as clinically indicated or until disease progression.
  * Percentage changes in total ctDNA (VAF), compared to baseline
Tumor uptake of [111In]-FPI-2107 | Within 56 days of administration
  • Tumor uptake of [111In]-FPI-2107 in selected regions of interest on SPECT/CT and/or planar images
Pharmacokinetics (PK) of [111In]-FPI-2107, and [225Ac]-FPI-2068, by measuring changes in clearance, AUC, Cmax, and half-life. | From first dose of investigation product until 56 days after the last dose of investigational product.
  • Determine the plasma concentrations and PK parameters of [111In]-FPI-2107, and [225Ac]-FPI-2068 and the effect of pre-dose administration of FPI-2053 on the plasma concentrations and PK parameters of [111In]-FPI-2107.
To assess the immunogenicity of [111In]-FPI-2107, [225Ac]-FPI-2068, and FPI-2053 | From first dose of investigation product until 56 days after the last dose of investigational product.
  • Presence of ADA for [111In]-FPI-2107, [225Ac]-FPI-2068, and FPI-2053

CONTACTS AND LOCATIONS:
Locations (15):
- United States (11):
  - Research Site, Irvine, California
  - Research Site, Palo Alto, California
  - Research Site, Santa Monica, California
  - Research Site, Chicago, Illinois
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Cleveland, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Houston, Texas
  - Research Site, Seattle, Washington
- Canada (4):
  - Research Site, Edmonton, Alberta
  - Research Site, Halifax, Nova Scotia
  - Research Site, Montreal, Quebec
  - Research Site, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/